University of Pennsylvania Institutional Review Board 3800 Spruce St., First Floor Suite 151 Philadelphia, PA 19104 Ph: 215-573-2540 (Federalwide Assurance # 00004028)

11-Apr-2019

Vera Krymskaya Attn: Sheila Pierson

spierson@pennmedicine.upenn.edu krymskay@mail.med.upenn.edu

PRINCIPAL INVESTIGATOR: Vera Krymskaya

TITLE : Research in Multicentric Castleman Disease

SPONSORING AGENCY : No Sponsor Number

PROTOCOL # : 823546 REVIEW BOARD : IRB #7

## Dear Dr. Krymskaya:

The above-referenced protocol received final review on 10-Apr-2019. As instructed, the project was closed. The protocol file will be archived according to University policies.

If you have any questions about the information in this letter, please contact the IRB administrative staff. Contact information is available at our website: http://www.upenn.edu/IRB/directory.

Thank you for your cooperation.

Sincerely,

Renee Digitally signed by Renee Crews
Date: 2019.04.15
13:55:02 -04'00'
IRB Administrator